CLINICAL TRIAL: NCT06483074
Title: Empagliflozin on Residual Kidney Function in Incident Peritoneal Dialysis Patients: a Pilot Randomized Controlled Trial
Brief Title: Empagliflozin on Residual Kidney Function in Incident Peritoneal Dialysis Patients
Acronym: EMPIRIC-PD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheuk-Chun SZETO, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CREC 2024.090-T
Record Dates: First submitted 2024-06-23; First posted 2024-07-01 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: End Stage Renal Disease on Dialysis; Peritoneal Dialysis Complication; Sodium-glucose Cotransporter-2 Inhibitor; Residual Kidney Function
MeSH Terms: interventions — empagliflozin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Active Comparator): Patients randomized to intervention group will receive oral empagliflozin 10mg daily on top of optimized dose of RAAS inhibitor for 6 months
  Interventions: Drug: Empagliflozin 10 MG
- Control group (No Intervention): Patients randomized to control group will receive optimized dose of RAAS inhibitor for 6 months

INTERVENTIONS:
Drug: Empagliflozin 10 MG — empagliflozin oral 10mg daily for 6 months
  Other Names: Jardiance 10mg daily
  Arms: Intervention group

SUMMARY:
Empagliflozin, a new class of diabetes medication, has demonstrated a reduction in renal function decline among patients with chronic kidney disease, regardless of their diabetes status. However, all previous studies excluded dialysis patients. Patients starting dialysis may still produce a certain amount of urine. Importantly, patients with better preserved residual kidney function tend to have better control of blood pressure and volume status, improved nutrition status, higher quality of life and reduced mortality rate.

The purpose of this study is to learn about the safety of empagliflozin in patients on peritoneal dialysis, in preparation for a future large clinical trial. Participants who newly initiate peritoneal dialysis will be randomly allocated to either empagliflozin on top of standard of care, or standard of care alone. Over a follow-up period of six months, the investigators will collect information on urine volume, blood pressure and glucose control. Safety, tolerability and drug compliance of empagliflozin will also be evaluated. If empagliflozin is found to be safe and well tolerated in patients on peritoneal dialysis, further large-scale randomized controlled trial may be conducted to evaluate its impact on residual kidney function and other relevant clinical outcomes.

DETAILED DESCRIPTION:
Diabetes is the leading cause of end stage kidney disease in developed countries. Peritoneal dialysis (PD) is a home-based and cost-effective modality of kidney placement therapy. Maintenance of residual kidney function (RKF) is one of the most crucial objectives to improve outcomes of PD patients. Observational studies showed that residual urine volume or residual glomerular filtration rate (GFR), but not peritoneal creatinine clearance, independently predicted patient survival. This benefit is likely attributed to better volume control, improved nutritional status, preserved endocrine function and enhanced clearance of uremic toxins in the presence of RKF. However, current therapeutic strategies to preserve RKF were most limited to the use of renin-angiotensin-aldosterone system (RAAS) inhibitors and biocompatible PD solutions.

Hong Kong adopted the 'PD-first' policy since 1985, and has the highest proportion of PD patients in the world. Inadequate dialysis, which is directly related to the loss of RKF, is the second most common reason for a permanent transfer to hemodialysis among PD patients. Sodium-glucose cotransporter-2 (SGLT-2) inhibitors have been shown to reduce albuminuria and delay progression of chronic kidney disease even in patients with advanced stages of kidney disease. It is postulated that the renoprotective effect of SGLT-2 inhibitors may be extended to dialysis population since a considerable proportion of patients still have urine output. SGLT2 inhibitors may potentially attenuate GFR decline in PD patients because heavy proteinuria independently predicted decline in residual GFR and onset of anuria. Moreover, preclinical studies suggested that empagliflozin reduced inflammation and oxidative stress by decreasing proinflammatory cytokines, inducing expression of anti-inflammatory M2 phenotype of macrophages, and antagonizing the effect of advanced glycation products. This beneficial effect may be particularly relevant to PD patients, where subclinical inflammation is common and inversely correlated with RKF.

Despite the potential promising effect of SGLT2-inhibitors in RKF in PD patients, dialysis patients were excluded in previous randomized controlled trials. In the present study, the investigators hypothesize that oral empagliflozin in addition to RAAS inhibitor, compared to RAAS inhibitor alone, better preserves RKF in patients newly started on PD. After a run-in period of 6 to 8 weeks where the dose of RAAS inhibitors are uptitrated to maximally tolerated dose, 48 incident PD patients will be randomized to empagliflozin or control (no empagliflozin) for a total of 6 months. This study aims to explore the feasibility of conducting a full-scale, adequately powered randomized controlled trial that investigates the effect of empagliflozin on RKF in incident PD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Incident PD patients within 90 days of Tenckhoff catheter insertion
2. Age 18-75 years old
3. Patient with or without history of Type 2 diabetes
4. Residual GFR (defined as the average of 24-hour urinary urea and creatinine clearances) > 2ml/min/1.73m2 AND urine volume > 400ml per day
5. Patients who are willing to provide written informed consent

Exclusion Criteria:

1. Patients with history of hemodialysis (≥ 3 months) or renal transplant
2. Life expectancy <6 months
3. Prior use of any type of SGLT2 inhibitors within 1 month before screening visit
4. Poorly controlled diabetes with HBA1c >11%
5. Type 1 diabetes
6. History of any active malignancy within 5 years (except curatively resected basal cell or squamous cell skin cancers)
7. Peritonitis within 4 weeks
8. Ketoacidosis within 5 years
9. Known hypersensitivity to empagliflozin or other SGLT2 inhibitors
10. Any active acute or chronic physical or mental conditions that, in the opinion of the investigator, might interfere with the compliance of participants to or the performance of this study
11. Participation in any clinical trial or use of any investigational medicinal product 1 month before screening visit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | During randomization
  Number of patients who are randomized each month following the run-in period
Medication adherence | 6 months
  Proportion of prescribed empagliflozin that are taken by the patients (pill counting will be done by investigators at each follow up)
Retention rate | 6 months
  Proportion of patients who have completed the whole study among patients that are randomized

SECONDARY OUTCOMES:
Slope of residual GFR | 6 months
  Residual GFR is calculated as the arithmetic mean of 24-hour urinary urea and creatinine clearances
Time to anuria | 6 months
  Anuria is defined as urine volume <100ml per day
Difference in residual urine volume | Month 0, 2, 4, 6
  Residual urine volume is measured by 24-hour urine collection
Difference in volume of overhydration | Month 0, 2, 4, 6
  Volume of overhydration is measured by a validated multi-frequency bioimpedance spectroscopy
Difference in plasma N-terminal pro-brain type natriuretic peptide | Month 0, 2, 4, 6
  Indicator for left ventricular dysfunction
Difference in systolic blood pressure | Month 0, 2, 4, 6
  Office blood pressure will be measured according to standardized protocol. The average of three consecutive measurements by an automated device will be recorded.
Difference in volume of ultrafiltration per day | Month 0, 1, 2, 4, 6
  The volume of fluid removed from patient by peritoneal dialysis each day
Incidence of urinary tract infection | 6 months
  Proportion of patients who have symptoms consistent with urinary tract infection and organisms identified by urine culture
Incidence of genital tract infection | 6 months
  Proportion of patients who are symptomatic and require antibiotic or anti-fungal treatment
Incidence of ketoacidosis | 6 months
  Proportion of patients who have serum pH <7.3 and elevated serum beta hydroxybutyrate ≥3.0 mmol/L
Incidence of lower limb amputation | 6 months
  Proportion of patients who require lower limb amputation by operation that is not secondary to trauma
Incidence of severe hypoglycemia | 6 months
  Proportion of patients who have hypoglycemia requiring third party assistance

OTHER OUTCOMES:
Change in peritoneal solute transfer rate | Month 0, 6
  This is measured by dialysate-to-plasma creatinine ratio in a standard peritoneal equilibration test (PET)
Difference in frailty status by Clinical Frailty Scale | Month 0, 6
  Clinical Frailty Scale is 9-point scale which is used to quantify the frailty and functional status of dialysis patients. A higher score indicates greater degree of frailty.
Difference in frailty status by Fried frailty phenotype | Month 0, 6
  Fried phenotype consists of five criteria which include both patient-reported domains and objective assessments. Subjects are considered to be frail if they meet three or more criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Jack KC Ng, FRCP, Principal Investigator — Chinese University of Hong Kong; Cheuk Chun Szeto, MD, FRCP, Study Director — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No